CLINICAL TRIAL: NCT04126512
Title: Effect of the Timing of Surgical PDA Ligation on Neonatal Outcomes: a Bicentric Retrospective Observational Study.
Brief Title: Timing of Surgical PDA Ligation and Neonatal Outcomes
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Silvia Martini, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: PDA-lig-SO-CAM
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Patent Ductus Arteriosus; Patent Ductus Arteriosus - Delayed Closure; Patent Ductus Arteriosus After Premature Birth
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bedside ligation: Infants admitted to St. Orsola-Malpighi Hospital (SOM) NICU had their PDA ligated at bedside, with a timing of surgery dependent on the time schedule of the surgeons and anaesthesiologists.
  Interventions: Other: PDA ligation
- Referred to specialist paediatric cardiac surgery centre: Due to the unavailability of local cardiac surgery, infants admitted to the Cambridge University Hospital (CUH) NICU were referred to specialist paediatric cardiac surgical centres, where PDA ligation was performed. In these cases, the surgical timing depended on both bed availability at the referral centre and the availability of the neonatal transfer team.
  Interventions: Other: PDA ligation

INTERVENTIONS:
Other: PDA ligation — PDA ligation was performed at bedside, if a local cardiac surgery team was available, or in the case this service was not available, infants were referred to off-site specialist paediatric cardiac surgical services, where PDA ligation was performed.

SUMMARY:
Patent ductus arteriosus (PDA) is common among very preterm infants. If pharmacological closure is ineffective or contraindicated, surgical ligation may be required. Access to cardiothoracic surgery may influence the timing of ligation, with possible long-term clinical effects. This study protocol aims to assess the impact of different surgical management of PDA (bedside surgery vs. referral to a cardiac surgery centre) on ligation timing and neonatal clinical outcomes in two tertiary Neonatal Intensive Care Units.

Infants born at St. Orsola-Malpighi University Hospital, Bologna, Italy (group 1, bedside ligation) and Cambridge University Hospital, Cambridge, UK (group 2, referred to an off-site specialist paediatric cardiac surgical centre) who underwent PDA ligation between 2007 and 2018 will be included in this retrospective cohort study if fulfilling the following criteria: gestational age (GA) <32 weeks, birth weight (BW) <1500 g, inborn, absence of major malformation or congenital heart disease. Neonatal clinical outcomes will be collected and compared between the 2 groups.

DETAILED DESCRIPTION:
Patent ductus arteriosus (PDA) is a common condition among preterm infants, with an estimated incidence of 60% in extremely low birth weight infants (ELBW). Several factors, such as the relative oxygen hyposensitivity and increased sensitivity to prostaglandins of the immature tissues and the scarceness of ductal medial muscles, contribute to the patency of arterial duct in prematurely born neonates; as a consequence, the rate of spontaneous closure is inversely related to gestational age (GA) Over the past two decades, the persistence of a significant systemic-to-pulmonary shunt through the PDA has been associated with a higher incidence of adverse clinical outcomes, including acute pulmonary morbidities and bronchopulmonary dysplasia (BPD), intraventricular haemorrhage (IVH), necrotizing enterocolitis (NEC), feeding intolerance and increased mortality rates.

The management of PDA in very preterm infants first includes supportive therapy (e.g., restricted fluid intake, diuretics, increasing end-expiratory pressure) and targeted pharmacologic treatment with cyclooxygenase inhibitors (i.e., ibuprofen, indomethacin, acetaminophen) or paracetamol if spontaneous closure does not occur. However, when pharmacological closure is ineffective or contraindicated and the neonate requires extensive respiratory support, surgical ligation may be required. PDA ligation can be performed on-site, either at the infants' bedside or in the operation room, or off-site, if a paediatric cardiac surgery team is not available locally. By favouring one approach over the other, the setting may also contribute to influence the timing for PDA ligation. To date, literature comparing the effects of early vs. delayed PDA ligation on the main neonatal morbidities has led to contrasting results; hence, the optimal timing of surgical PDA closure remains a matter of debate among neonatologists.

This study aims to assess whether a different management of surgical PDA closure (on-site bedside ligation vs. referral to an off-site specialist paediatric cardiac surgical centre) may influence the timing of the intervention and the main neurological, respiratory and gastrointestinal clinical outcomes in very low birth weight (VLBW) preterm infants from two tertiary Neonatal Intensive Care Units with different paediatric cardiac surgery capabilities. Postoperative complications, mortality rates and the length of hospital stay will be also evaluated as secondary outcomes.

Methods Preterm infants <32 weeks' gestation born at the Neonatal Intensive Care Unit (NICU) of Cambridge University Hospital (CUH, Cambridge, UK) and of St. Orsola-Malpighi Hospital (SOM, Bologna, Italy) between January 1st, 2007 and June 30th, 2018 will be included in this retrospective study if, due to failed or contraindicated medical therapy, underwent surgical closure of PDA, judged hemodynamically significant (hsPDA) either on a clinical (hypotension, ventilator dependence, heart failure symptoms) or echocardiographic basis (left atrial/aortic root ratio >1.5, pulsatile left-to-right shunt and/or mean velocity in the left pulmonary artery >0.6 m/s). The presence of major congenital malformations, including congenital heart disease, was considered an exclusion criterion.

Echo-Doppler studies of each patient will be reviewed, and the following parameters from the latest pre-operative scan were will be recorded: PDA size and shunt characteristics (direction and pattern); left atrial to aortic root ratio; evidence of reversed end-diastolic flow in the descending aorta and/or in the middle or anterior cerebral artery (when evaluated). Contraindications and adverse effects of pharmacological treatment will be also reviewed. Failure of pharmacological treatment is defined by PDA persistency after at least two full pharmacological courses.

Neonatal characteristics and the following pre- and peri-operative data will be recorded: echocardiographic PDA characteristics, PDA management (supportive or pharmacological treatment, related adverse effects, rates of responsiveness and recurrence), post-conceptional age, days of life and weight at surgical intervention.

Neonatal outcomes include mortality rates, IVH, periventricular leukomalacia (PVL), NEC, sepsis (defined as relevant symptoms with positive blood culture and/or C reactive protein >25 mg/L and >5 days of antibiotic treatment), retinopathy of prematurity (ROP, any grade) and BPD (defined as any requirement for supplemental oxygen and/or positive-pressure respiratory support at 36 weeks' post-conceptional age). Length of hospital stay, time needed to achieve full enteral feeding, total duration of mechanical ventilation and the rate of supplemental oxygen need at hospital discharge will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32 weeks' gestation
* Surgical PDA ligation

Exclusion Criteria:

* Major congenital malformations
* Congenital heart disease

Ages: 1 Day to 6 Months | Sex: All
Age Groups: Child
Study Population: Infants born at the Neonatal Intensive Care Unit (NICU) of Cambridge University Hospital (CUH, Cambridge, UK) and of St. Orsola-Malpighi Hospital (SOM, Bologna, Italy) between 01/01/2007 and 30/06/2018
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PDA ligation timing | From birth up to hospital discharge (average period: 6 months)
  Days of life at PDA ligation in SOM group compared to the CUH group
Mortality | From birth up to hospital discharge (average period: 6 months)
  Any decrease in the mortality rate in the SOM group compared to the CUH group
Bronchopulmonary dysplasia | 36 weeks' post-conceptional age
  Any decrease in the rate of bronchopulmonary dysplasia in the SOM group compared to the CUH group

SECONDARY OUTCOMES:
Intraventricular haemorrhage (IVH) | From birth up to hospital discharge (average period: 6 months)
  Any decrease in the incidence of IVH in SOM group compared to the CUH group
Periventricular leukomalacia (PVL) | From birth up to hospital discharge (average period: 6 months)
  Any decrease in the incidence of PVL in SOM group compared to the CUH group
Necrotizing enterocolitis (NEC) | From birth up to hospital discharge (average period: 6 months)
  Any decrease in the incidence of NEC in SOM group compared to the CUH group
Retinopathy of prematurity (ROP) | From birth up to hospital discharge (average period: 6 months)
  Any decrease in the incidence of ROP in SOM group compared to the CUH group
Oxygen need at discharge | Hospital discharge (average age: 6 months of life)
  Any decrease in the rate of oxygen need at discharge in SOM group compared to the CUH group
Length of hospital stay | Hospital discharge (average age: 6 months of life)
  Duration of hospitalization in the SOM group compared to the CUH group
Time to achieve full enteral feeding | From birth up to hospital discharge (average period: 6 months)
  Time needed to achieve full enteral feeding in the SOM group compared to the CUH group
Duration of mechanical ventilation | From birth up to hospital discharge (average period: 6 months)
  Days spent on mechanical ventilation in the SOM group compared to the CUH group

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Martini, MD, Principal Investigator — Sant'Orsola-Malpighi University Hospital
Locations (2):
- S. Orsola-Malpighi University Hospital, Bologna, Emilia-Romagna, Italy
- The Rosie Hospital, Cambridge University Hospitals, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No